CLINICAL TRIAL: NCT01536847
Title: Glycaemic Response Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Reading Scientific Services Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: P11-09257
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Glycaemic Index; Glycaemic Response
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Test Drink (Placebo Comparator): Control drink
  Interventions: Other: Dietary Intervention
- Experimental Test Drink 1 (Experimental): Control drink containing ingredient 1
  Interventions: Other: Dietary Intervention
- Experimental Test Drink 2 (Experimental): Control drink containing ingredient 2
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — 300 ml of liquid food product
  Arms: Control Test Drink
Other: Dietary Intervention — 300 mL of liquid food product
  Arms: Experimental Test Drink 1
Other: Dietary Intervention — 300 ml of liquid food product
  Arms: Experimental Test Drink 2

SUMMARY:
The purpose of this study is to assess whether added food ingredient(s) affect glycemic responses to a liquid meal tolerance test (LMTT).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (not less than 40% males or females
* Non-smoker
* Aged 18 to 55 years
* Have a body mass index between 18.5 to 29.99 kg/m2
* Healthy, non-diabetic, no gastric bypass surgery
* Having a fasting plasma glucose (finger stick) <100 mg/dl (<5.5 mmol/L)
* Willing and able to provide written informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Glycaemic index of experimental test food using capillary blood | 0-120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Suzana Louth, Dr, Principal Investigator — RSSL